CLINICAL TRIAL: NCT04412551
Title: Lung Ultrasound for Assessment of Patients With Moderate to Severe Covid-19
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Maria Hårdstedt, Dr. Maria Hårdstedt, PhD, Specialist Internal Medicine, Dalarna County Council, Sweden
Other Study IDs: LUS-Covid001
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Corona Virus Infection; Virus Diseases; Coronaviridae Infections
Keywords: ultrasonography; lung ultrasound; covid-19; ARDS
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; Coronaviridae Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will describe lung ultrasound (LUS) findings over time in hospitalized patients with moderate to severe Covid-19 lung disease. Our primary aim is to investigate if lung ultrasound can identify and/or predict patients requiring mechanical ventilation. Another aim is to describe LUS findings associated with clinical findings and patient condition.

DETAILED DESCRIPTION:
Study patients with moderate to severe Covid-19 infection will be screened with lung ultrasound daily. Lung ultrasound will be assessed by LUS-score for acute respiratory distress syndrome (ARDS) (0-36 points, Bouhemad 2015). Findings of B-line artifacts and consolidations will be noted. In addition to LUS, clinical parameters from physical examination and laboratory tests will be collected. Participants wil be followed until either admission to intensive care unit (ICU) for mechanical ventilation or until clinical improvement. A group of patients with mild Covid-19 infection will be recruited and screened once as reference.

Apart from assessment with LUS, patients are managed according to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 confirmed by positive polymerase chain reaction (PCR)
* oxygen by mask or nasal prongs ≥ 4 l/min or high flow nasal cannula (HFNC) with fraction of inspired oxygen (FiO2) ≥ 30%
* age between 18-80 years
* informed consent

Exclusion Criteria:

* patients subject to treatment-limitation "no ICU"
* history of heart failure
* history of lung disease e.g.: pneumonectomy, pulmonary fibrosis or other interstitial lung disease, pleurodesis
* history of kidney failure requiring dialysis
* any reason making lung ultrasound or daily follow up impossible
* opposition to participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients with confirmed Covid-19 and oxygen therapy corresponding to stage 4-5 on the "Ordinal Scale for Clinical Improvement" of the World Health Organization.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of requirement of mechanical ventilation | 3 weeks
  Assessment of LUS-score or findings of consolidations correlated to requirement of mechanical ventilation on ICU

SECONDARY OUTCOMES:
Prediction of requirement of mechanical ventilation | 3 weeks
  Assessment if LUS-score or findings of consolidations is able to anticipate clinical deterioration with requirement of mechanical ventilation on ICU
Association of LUS to clinical parameters | 3 weeks
  Descriptive assessment of clinical parameters and LUS-score over time
Description of findings on LUS | 3 weeks
  Description of quality and distribution pattern of LUS-findings in patients with different severities of Covid-19

CONTACTS AND LOCATIONS:
Locations (1):
- Falun Hospital, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouhemad B, Mongodi S, Via G, Rouquette I. Ultrasound for "lung monitoring" of ventilated patients. Anesthesiology. 2015 Feb;122(2):437-47. doi: 10.1097/ALN.0000000000000558. No abstract available. PMID 25501898